CLINICAL TRIAL: NCT03453450
Title: Exploring Volunteers' Experiences in Health TAPESTRY, a Primary Care-Based Program
Brief Title: Exploring Volunteers' Experiences in Health TAPESTRY
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Red Cross (Other); David Braley (Unknown); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Other Study IDs: 4301
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-09

CONDITIONS: Volunteers
Keywords: Primary Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health TAPESTRY volunteers: Volunteers in a primary care setting connecting with Health TAPESTRY clients
- Health TAPESTRY Volunteer Coordinators: The coordinators of volunteers

SUMMARY:
This study is meant to evaluate the Health TAPESTRY volunteer program. The objective of this study is to explore volunteer experiences in Health TAPESTRY in terms of implementation and to understand how participation in Health TAPESTRY as a volunteer is related to compassion, self-reported physical activity, quality of life, and attitudes toward older adults.

DETAILED DESCRIPTION:
Health TAPESTRY aims to help people stay healthier for longer in the places where they live. As a person-focused, proactive approach, Health TAPESTRY incorporates trained community volunteers into the primary care team in a way that is seamless and complementary to the essential work that clinicians are undertaking each day. In the program, volunteers conduct home visits with older adult clients, complete questionnaires, and connect their clients to primary care and community resources. This study offers the opportunity to fill a major gap in the literature by investigating the experiences of volunteers within Health TAPESTRY and the effect on them of participation as an intervention in its own right.

Specifically, the study seeks to understand volunteers' experiences in the program and evaluate any effects that volunteering with the program has on the volunteers including with the volunteers health and wellness (specifically physical activity and quality of life), empathy, and attitudes toward older adults. The investigators will also look at how the volunteers patterns of compassion fatigue and compassion satisfaction might change throughout involvement in the program, and how that connects to volunteer demographic characteristics like age and gender, as well as other characteristics like empathy, how many home visits are conducted, and the initial motivation to volunteer with the program.

This program evaluation study will employ qualitative and quantitative data collection strategies including surveys, narratives written by volunteers, and volunteer focus groups.

ELIGIBILITY:
Must be a Health TAPESTRY Volunteer or Volunteer Coordinator. There are no further inclusion or exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants are drawn from the Health TAPESTRY volunteer pool. All Health TAPESTRY volunteers will be invited into the evaluation, however only those volunteers who choose to take part in the evaluative component of the program will be included in the analysis. Although we aim to include as many Health TAPESTRY volunteers as possible, an achievable target is set at half of the volunteers (approximately 17) in each of the 6 sites being involved in the research component.
  The Volunteer Coordinator (VC) in each site will also be invited to attend an interview. The day-to-day management of volunteers within each site is managed by a VC from the Canadian Red Cross. The VC is the first contact for volunteers, and also the primary conduit that connects volunteers with clients.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Volunteers' Experiences | 12 months
  Volunteers' and volunteer coordinators' perceptions about their experiences in Health TAPESTRY overall, and specifically in regards to their understanding of their role; the training that was offered and how it did or did not support them in carrying out their role effectively; the process of engagement in the program from onboarding through the volunteer coordination to conducting home visits with clients; and the perceived outcomes of volunteering, including the impact of volunteering on their own health and wellness. This will be collected through qualitative data: focus groups for volunteers and interviews for volunteer coordinators at the 12-month mark, and volunteer narratives which are written post-client-visits.

SECONDARY OUTCOMES:
Compassion satisfaction and compassion fatigue | Baseline, 3 month, 6 month, 9 month, 12 months
  The change in compassion over time during participation as a Health TAPESTRY volunteer will be measured via the Professional Quality of Life survey (ProQOL), which measures both compassion fatigue and compassion satisfaction through 30-items on 5-point scales ranging from "never" to "very often". Collected every 3 months for a 12 month period.
Physical Activity | Baseline, 12 months
  Volunteers' physical activity will be measured via the International Physical Activity Survey (IPAQ). Respondents indicate how many days in the past seven days, and for how many minutes, they have engaged in vigorous and moderate intensity activity and walking activity. Scores for vigorous and moderate intensity activity, and walking activity are calculated by multiplying the days by the number of minutes on one day by the metabolic equivalent of task (MET) value for the activity. The MET values used for vigorous and moderate intensity activity and walking are 8.0, 4.0, and 3.3 respectively. Collected at baseline and 12 months.
Quality of Life | Baseline, 12 months
  Volunteers' quality of life will be measured via the five-level EuroQol five-dimension (EQ-5D-5L). The EQ-5D-5L asks respondents to rate their current ability in five domains: mobility, self-care, usual activities, pain, and anxiety/depression, on a five-level scale. In addition, respondents are asked to rate their current health state on a scale from 0 ('worst health you can imagine') to 100 ('best health you can imagine'). A score from the five domains is calculated using a macro program and ranges from 0 to 1. Collected at baseline and 12 months.
Attitudes Toward Older Adults | Baseline, 12 months
  Volunteers' attitudes toward older adults will be measured via the UCLA Geriatric Attitudes Scale.This 14-item survey measures volunteers' attitudes of older adults on a 5-point scale ranging from "strongly disagree" to "strongly agree". Collected at baseline and 12 months.
Empathy | Baseline, 12 months
  Volunteer empathy will be measured via the Basic Empathy Scale (BES), a 20-item scale based on a two-factor model of empathy. It includes 9 items evaluating cognitive empathy and 11 items evaluating affective empathy. Participants are asked to respond to each item on a five-point scale ranging from "strongly disagree" to "strongly agree". With permission from the author, language on the BES was slightly altered to fit a North American audience. Collected at baseline and 12 months.
Reasons for Volunteering | Baseline
  A subscale of Clary & Snyder's Volunteerism Questionnaire, the Reasons for Volunteering sub-scale has 20-items and asks participants to respond to each item on a 7-point scale ranging from "not at all important/accurate for you" to "extremely important/accurate for you". Collected at baseline.
Outcomes of Volunteering | 12 Months
  A subscale of Clary & Snyder's Volunteerism Questionnaire, the Volunteering Outcomes sub-scale has 18 items, and primarily asks participants to respond to each item on a 7-point scale ranging from "strongly disagree" to "strongly agree". Collected at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Oliver, MSc,MD,CCFP, Principal Investigator — McMaster University; Dee Mangin, MBChB,DPH,FRN, Principal Investigator — McMaster University
Locations (1):
- David Braley Health Sciences Centre, McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No